CLINICAL TRIAL: NCT02999646
Title: Personalized and Cell-based Antitumor Immunization MVX-ONCO-1 in Advanced Head and Neck Squamous Cell Carcinoma. A Single Arm, Open Label, Multicenter Phase II Trial.
Brief Title: Personalized and Cell-based Antitumor Immunization MVX-ONCO-1 in Advanced HNSCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maxivax SA (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 11/16
Record Dates: First submitted 2016-12-19; First posted 2016-12-21 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma; cancer; HNSCC; immunotherapy; MVX-ONCO-1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Neoplasms

STUDY DESIGN:
Intervention Model Description: antitumor immunization MVX-ONCO-1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MVX-ONCO-1 (Experimental): MVX-ONCO-1 vaccine treatment once weekly starting on week 1 for 4 weeks followed by two additional treatments 2 weeks apart (total 6 treatments over 8 weeks). Each treatment consists of two macrocapsules containing the MVX-1 cell line and lethally irradiated autologous tumor cells.
  Interventions: Other: MVX-ONCO-1

INTERVENTIONS:
Other: MVX-ONCO-1 — Autologous cells: 1 vial containing 4x10^6 irradiated tumor cells Capsules: 2 biocompatible capsules loaded with 8x10^5 MVX-1 cells

SUMMARY:
The purpose of this trial is to determine the efficacy of the immunotherapy with MVX-ONCO-1 in patients with advanced head and neck squamous cell carcinoma. MVX-ONCO-1 consists of dead tumor cells from the patient itself and genetically modified cells within a capsule. The whole treatment takes 9 weeks. At weeks 1, 2, 3, 4, 6 and 8, the tumor cells are injected underneath the skin and two capsules are implanted for a week. At weeks 2, 3, 4, 5, 7 and 9 the capsules are removed again. The patients are then followed-up for 5 years.

DETAILED DESCRIPTION:
Patients with advanced HNSCC after platinum-based palliative chemotherapy have a poor prognosis, with no well-defined standard treatment and a survival between 6 to 9 months.

MVX-ONCO-1 is a patient specific, cell-based, active immunotherapy, where the patient's immune response to tumor cells is stimulated and/or increased by triggering an immune response against the patients' cancer cells.

Rationale for this trial is:

1. HNSCC: there is a clear medical need in this patient population,
2. Relapsing HNSCC often have accessible tumor tissue,
3. HNSCC is considered an immunogenic tumor.

This phase II study is a first step towards a potentially innovative immunotherapy for HNSCC.

MVX-ONCO-1 is composed of:

1. An immune-modulator (GM-CSF: granulocyte-macrophage colony stimulating factor) released from an immuno-protected, encapsulated, allogeneic, genetically modified cell line (MVX-1), and
2. Irradiated, autologous tumor cells as source of antigen.

Each treatment consists of two macrocapsules containing the MVX-1 cell line implanted subcutaneously and lethally irradiated autologous tumor cells injected subcutaneously. Eligible patients will receive a treatment once weekly starting on week 1 for 4 weeks followed by two additional treatments 2 weeks apart (total 6 treatments over 8 weeks). Each pair of macrocapsules is removed after 1 week, and the last implanted capsules are removed in week 9. The patients are then followed-up for 5 years.

The project has received funding from the European Union's Horizon 2020 research and innovation programme under grant agreement No 880194.

ELIGIBILITY:
Inclusion Criteria for pre-registration:

* Written informed consent according to ICH/GCP regulations before pre-registration
* Histologically confirmed diagnosis of head and neck squamous carcinoma (oral cavity, pharynx, larynx), Stage III/IV in recurrent or metastatic stage. Patients with local relapse for whom a curative treatment is available cannot be enrolled. Furthermore, all patients should have no other therapeutic option left.
* At least one line of prior anticancer therapy for recurrent or metastatic disease. Patients with locally advanced disease experiencing local relapse within 6 months of last dose of curative intended, platinum-based chemo-radiation with or without prior surgery can also be included.
* Primary tumor and/or metastasis amenable for partial/total surgery or tap
* Measurable or evaluable disease according to RECIST 1.1 criteria
* Patients age ≥ 18 years
* WHO performance status 0-2
* Adequate hematological values: neutrophils ≥1x10^9/L, platelets ≥70x10^9/L
* Adequate hepatic function: bilirubin ≤2 x ULN; AST and ALT and AP ≤2.5 x ULN (except for patients with liver metastasis: ≤5 x ULN)
* Adequate renal function (creatinine clearance >40mL/min/1.73m^2, calculated according to the corrected formula of Cockcroft-Gault
* Women with child-bearing potential are using effective contraception, are not pregnant and agree not to become pregnant after pre-registration, during trial treatment and during the 6 months thereafter. A negative blood pregnancy test before inclusion into the trial is required for all women with child-bearing potential
* Men agree not to father a child during trial treatment and during 6 months thereafter

Exclusion Criteria for pre-registration:

* Known or suspected CNS metastases or active leptomeningeal disease
* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years from registration with the exception of T1-2 prostate cancer Gleason score <6 (PSA<10 ng/mL), adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer
* Participated in any other investigational study or received an experimental therapeutic procedure considered to interfere with the study in the 4 preceding weeks of the pre-registration
* Concomitant use of other anti-cancer drugs
* Planned radiotherapy (other than symptom control)
* Severe or uncontrolled cardiovascular disease uncontrolled hypertension (sustained systolic blood pressure > 150 mm Hg and/or diastolic > 100 mm Hg despite antihypertensive therapy)
* History of cerebrovascular accident or intracranial hemorrhage within 6 months prior to pre-registration
* Any history of HIV
* Known history of HTLV-1, HTLV-2, or active chronic Hepatitis C or Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (iv) antimicrobial treatment
* Known severe allergy to reagents in the study product (MVX-ONCO-1)
* Systemic disease other than cancer that is not controlled by approved medication
* Patient with active autoimmune disease
* Chronic immunosuppressive treatment exceeding 20 mg/day of prednisone or an equivalent corticosteroid. Note: In acute situations prednison exceeding 20mg/day or equivalent(day is allowed during 7 days)
* Women who are pregnant or breast feeding
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications

Inclusion criteria for registration:

* Primary tumor and/or metastasis amenable for partial/total surgery or tap and subsequent cell harvest > 26x10^6 cells
* Measurable or evaluable disease according to RECIST 1.1 criteria
* WHO performance status 0-2
* Baseline QoL forms have been completed
* Adequate hematological values: neutrophils ≥1x10^9/L, platelets ≥70x10^9/L
* Adequate hepatic function: bilirubin ≤2 x ULN; AST and ALT and AP ≤ 2.5 x ULN (except for patients with liver metastasis: ≤5 x ULN)
* Adequate renal function (creatinine clearance >40 mL/min/1.73m^2, calculated according to the corrected formula of Cockcroft-Gault
* Women with child-bearing potential are using effective contraception, are not pregnant or lactating and agree not to become pregnant after registration, during trial treatment, and during the 6 months thereafter. A negative blood pregnancy

Exclusion criteria for registration:

* Known or suspected CNS metastases or active leptomeningeal disease
* Concomitant use of other anti-cancer drugs
* Planned radiotherapy (other than symptom control)
* Any one full cycle of anti-cancer chemotherapy treatment in the 3 preceding weeks of the registration
* Systemic disease other than cancer, that is not controlled by approved medication
* Chronic immunosuppressive treatment exceeding 20 mg/day of prednisone or an equivalent corticosteroid. Note: In acute situations prednisone exceeding 20 mg/day or equivalent is allowed during 7 days
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Overall Survival at 26 weeks (OS) | at 26 weeks from registration
  The primary endpoint of the trial is Overall Survival (OS) at 26 weeks defined as percentage of patients alive 26 weeks from registration. Patients who are lost to follow-up with a date they were last known to be alive less than 26 weeks after registration will be counted as failures for this endpoint.

SECONDARY OUTCOMES:
Time to subsequent therapy (TST) | assessed within 5 years
  defined as time from registration until documented start of subsequent therapy. Patients who did not start a subsequent therapy will be censored at the last date they were known to be alive
Duration of response (DOR) | assessed within 5 years
  defined as time from the date when a patient first meets the criteria for complete response (CR) or partial response (PR) until documented radiologic progression, relapse, or death due to disease progression, whichever occurs first. Patients not having an event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of their last tumor assessment showing non-progression before starting a new treatment. DOR will only be analyzed in the subgroup of patients achieving CR or PR during trial treatment based on RECIST 1.1.
Objective response rate (ORR) | at 6, 13, 26, 39 and 52 weeks
  defined as the proportion of patients having CR or PR at the respective time point after registration plus/minus 1 week at week 6, 13, 26, and plus/minus 2 weeks at week 39 and 52 after registration.
  The response rate will be analyzed based on RECIST 1.1. CR and PR will only be counted if the response is confirmed at least 4 weeks later
Disease control rate (DCR) | at 6, 13, 26, 39 and 52 weeks
  defined as the proportion of patients having CR, PR, or stable disease (SD) at the respective time point after registration plus/minus 1 week at week 6, 13, 26, and plus/minus 2 weeks at week 39 and 52 after registration. The disease control rate will be analyzed based on RECIST 1.1. CR and PR will only be counted if the response is confirmed at least 4 weeks later.
Best overall response | assessed within 5 years
  defined as best response achieved at any time during or after the trial treatment before starting a new anticancer treatment. Best overall response will be analyzed based on RECIST 1.1. CR and PR will only be counted if the response is confirmed at least 4 weeks later.
Objective response according to iRECIST (iOR) | at 6, 13, 26, 39 and 52 weeks
  defined as any complete response (CR/iCR) or partial response (PR/iPR) according to RECIST1.1 or iRECIST criteria achieved before new anti-cancer treatment is given. Any patient with CR/iCR or PR/iPR as best observed response under trial treatment will be considered as a success; otherwise they will be considered as a failure. Patients without any tumor assessment or with non-evaluable response (NE) under trial treatment will be considered as failures for this endpoint.
Progression Free Survival (PFS) | assessed within 5 years
  defined as the time from registration until progression according to RECIST 1.1 or death from any cause, whichever occurs first. Patients not having an event at the time of analysis and patients starting a new anticancer therapy in the absence of an event will be censored at the date of their last tumor assessment showing non-progression before starting a new treatment.
Progression-free survival according to iRECIST (iPFS) | assessed within 5 years
  defined as the time from registration until disease progression according to iRECIST criteria (iPD) or death due to any reason, whichever occurs first.
PFS at 6, 13, 26, 39, and 52 weeks | at 6, 13, 26, 39, and 52 weeks
  will be estimated using the Kaplan-Meier estimator for PFS at the respective time point after registration plus/minus 1 week at week 6, 13, 26, and plus/minus 2 weeks at week 39 and 52 after registration.
OS | assessed within 5 years
  defined as time from registration until death from any cause. Patients which are still alive will be censored at the date they were last known to be alive.
PFS under the first subsequent treatment | assessed within 5 years
  defined as the time from start of the first subsequence treatment until progression according to RECIST 1.1 or death from any cause, whichever occurs first. Patients not having an event at the time of analysis and patients starting next line of anticancer therapy in the absence of an event will be censored at the date of their last tumor assessment showing non-progression before starting new treatment.
Adverse and serious adverse events | assessed within 5 years
  All adverse events (AE) will be assessed according to NCI CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Michielin, Prof, Study Chair — CHUV Lausanne
Locations (4):
- Switzerland (4):
  - HUG Hôpitaux Universitaires Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez E, Vernet R, Urwyler M, Von Rohr O, Charrier E, Belkouch MC, Saingier V, Courtout F, DeVito C, Ancrenaz V, Dulguerov N, Karenovics W, Grogg J, Renaux J, Gobat K, Muller G, Brezina T, Rordorf T, Joerger M, Michielin O, Villard J, Mach N. Overall survival of recurrent/metastatic head & neck squamous cell carcinoma patients progressing after >/= 1 line of systemic therapy, treated with MVX-ONCO-1, a novel, first in class cell encapsulation-based immunotherapy: results of SAKK 11/16, a phase IIa trial. Exp Hematol Oncol. 2025 Aug 31;14(1):113. doi: 10.1186/s40164-025-00703-x. PMID 40887652